CLINICAL TRIAL: NCT00977457
Title: Pre-Surgical EPS Biomarkers as Predictors of Biochemical Recurrence
Brief Title: Genetic Testing in Predicting Biomarkers of Recurrence in Patients With Prostate Cancer Undergoing Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06072; P30CA033572 (NIH); CHNMC-06072; CDR0000644208 (Registry Identifier: NCI PDQ); 5R01CA102521 (NIH); NCI-2011-00980 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-09-12; First posted 2009-09-15 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — DNA Methylation; Gene Expression Profiling; Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (specimen collection) (Experimental): Patients receive prostatic massage and undergo a digital rectal examination. Laboratory assessments are performed and blood samples are collected for molecular biology testing. On the day of the scheduled prostatectomy, a second blood collection is performed prior to surgery.
  Interventions: Genetic: DNA analysis; Genetic: DNA methylation analysis; Genetic: RNA analysis; Genetic: gene expression analysis; Genetic: polymerase chain reaction; Other: diagnostic laboratory biomarker analysis; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Genetic: DNA analysis — Performed on Post-massage urine (PMU) and/or expressed prostatic secretions (EPS) samples obtained at the time of surgery
Genetic: DNA methylation analysis — Performed on Post-massage urine (PMU) and/or expressed prostatic secretions (EPS) samples obtained at the time of surgery
Genetic: RNA analysis — Performed on Post-massage urine (PMU) and/or expressed prostatic secretions (EPS) samples obtained at the time of surgery
Genetic: gene expression analysis — Performed on Post-massage urine (PMU) and/or expressed prostatic secretions (EPS) samples obtained at the time of surgery
Genetic: polymerase chain reaction — Performed on Post-massage urine (PMU) and/or expressed prostatic secretions (EPS) samples obtained at the time of surgery
Other: diagnostic laboratory biomarker analysis — Performed on Post-massage urine (PMU) and/or expressed prostatic secretions (EPS) samples obtained at the time of surgery
Procedure: therapeutic conventional surgery
  Other Names: Undergo robotic prostatectomy or cystoprostatectomy

SUMMARY:
This trial studies the side effects and best way to perform genetic testing in predicting biomarkers of recurrence in patients with prostate cancer undergoing surgery. Collecting and storing samples of tissue, blood, and other body fluids from patients to test in the laboratory and collecting information about the patient's health and treatment may help doctors learn more about cancer and help predict the recurrence of prostate cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To explore the performance of these models in predicting the likelihood of biochemical recurrence (BCR).

SECONDARY OBJECTIVES: I. To explore the performance of these models in predicting upgrading and upstaging prior to surgery. II. To explore the performance of these models in improving risk stratification among patients eligible for active surveillance. III. To determine whether prostatic massage or surgery raises the count of circulating tumor cells (CTC) in post-digital rectal exam (DRE) blood specimens.

OUTLINE: Patients receive prostatic massage and undergo a digital rectal exam (DRE). Laboratory assessments are performed and blood samples are collected for molecular biology testing. On the day of the scheduled prostatectomy, a second blood collection is performed prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

- All men undergoing robotic prostatectomy or cystoprostatectomy at City of Hope will be eligible for the study

Exclusion Criteria:

- Men who undergo neoadjuvant treatment with Androgen Deprivation Therapy (ADT) or salvage prostatectomy including those who have had brachytherapy will be excluded

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1045 (Actual)
Dates: Start 2007-11-26 (Actual); Primary Completion 2016-07-13 (Actual); Study Completion 2026-07-08 (Estimated)

PRIMARY OUTCOMES:
Performance of these models in predicting the likelihood of BCR | Visit 2 (intraoperative setting)
  Logistic regression and artificial neural networks will be used.

SECONDARY OUTCOMES:
Comparison of the performance in these models in predicting upgrading and upstaging prior to surgery | Visit 2 (intraoperative setting)
  Logistic regression and artificial neural networks will be used.
Comparison of the performance of these models in improving risk stratification among patients eligible for active surveillance | Visit 2 (intraoperative setting)
  Logistic regression and artificial neural networks will be used.
Determination whether prostatic massage or surgery raises the count of circulating tumor cells (CTCs) in post-DRE blood specimens | Visit 2 (intraoperative setting)
  Logistic regression and artificial neural networks will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Steven S. Smith, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States